CLINICAL TRIAL: NCT04212897
Title: Therapeutic Benefits of Music for Parkinson's Disease: a fNIRS Study Protocol for Controlled Trial
Brief Title: fNIRS Studies of Music Intervention of Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Dalian Medical University (Other)
Collaborators: Dalian University of Technology (Unknown); University of California, Irvine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PJ-KY-2019-123
Record Dates: First submitted 2019-12-17; First posted 2019-12-30 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Music Therapy; fNIRS; Controlled Trials; Explicit & Implicit Timing; Motor Control; Synchronous finger tapping
MeSH Terms: conditions — Parkinson Disease | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients and the outcomes assessor are blinded in this study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Therapy (Experimental): This group will be asked to practice a rhythmic auditory SFT intervention task at home.
  Interventions: Other: Music Therapy
- No Music Therapy (No Intervention): This group will not engage in an intervention task at home and will be asked to continue their normal daily routine.

INTERVENTIONS:
Other: Music Therapy — Participants in the intervention arm will be asked to practice a rhythmic auditory synchronous finger tapping intervention task at home for a total of 25 minutes split between two ten-minute sets with a five-minute break between the sets every day for 8-weeks. During training sessions participants must listen to the instrumental of a pre-selected well-known Chinese melody, "Moonlight over the Lotus Pond" by Phoenix Legend, whose melody duration is 259s. This song was selected for its strong beat and familiarity to the participants. Participants must follow the beats of the melody and tap their right index finger simultaneously to the beats. A visual cue will be displayed to indicate the beats, identical to the one in the assessment. The training session will be conducted once daily after patients have taken their medication. Participants' primary caretaker will be asked to monitor and record completion of sessions.
  Arms: Music Therapy

SUMMARY:
Functional near-infrared spectroscopy (fNIRS) will be used to monitor neuronal activities and connectivity to elucidate the correlation between physiological changes within the brain and the benefits of music therapy for patients afflicted with Parkinson's disease (PD). This study will report on the changes in neural activities as a result of music intervention in PD.

DETAILED DESCRIPTION:
Music therapy improves neuronal activity and connectivity of healthy persons and patients with clinical symptoms of neurological diseases like Parkinson's Disease. Despite the plethora of publications that have reported the positive effects of music interventions, little is known about how music improves neuronal activity and connectivity in afflicted patients. In this study, the investigators will use functional near-infrared spectroscopy (fNIRS) to measure oxygenated- (HbO2), deoxygenated- hemoglobin (HbR), and total hemoglobin activation in various parts of the cortex. The fNIRS measurement, in conjunction with the Unified Parkinson's Disease Rating Scale (UPDRS), n-back task, and the Montreal Cognitive Assessment (MoCA), will be performed at baseline, week 4 (during), week 8 (post), and week 12 (retention) of the study. The 8-week long intervention will include a daily 25-minute synchronous finger tapping (SFT) intervention (two sets of ten-minute sessions with a five-minute break in between sets) with a pre-selected well-known rhythmical song. The total anticipated number of participants is 150 and the participants will be split into two groups: an intervention group and a control group. Data collected from the two PD groups will be compared to baseline performances from healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-80 years old, both genders, and right handed;
* Clinical diagnosis of idiopathic PD according to the 2015 Movement Disorder Society (MDS) Clinical Diagnostic Criteria for Parkinson's Disease;
* Rated as stage I to II on the Hoehn and Yahr scale;
* Scores greater than 21 points on the Montreal Cognitive Assessment (MoCA);
* Maintain a stable dosing of anti-PD or deep-brain stimulation (DBS) treatment throughout the duration of the study;
* Able to travel to and participate in the data collection process.

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria;
* Presence of significant hearing or visual impairments;
* Extensive previous musical training;
* A history of any other neurological condition (i.e. Alzheimer's disease, epilepsy, stroke) or psychiatric disorders (i.e. major depression, psychoses).

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change from Functional Near-infrared Spectroscopy from baseline | Week 0 (baseline), week 4 (during), week 8 (end), and week 12 (follow-up)
  An ETG-4000 fNIRS system will be used to measure hemoglobin (HBO2) levels in the participant as they perform finger motor control timing assessments. A change, specifically a reduction of HBO2 activation, from baseline measurements indicates reduced cortical activation and suggests improved PD-related symptoms.
Change in Synchronous Finger Motor Control Timing Abilities from baseline | Week 0 (baseline), week 4 (during), week 8 (end), and week 12 (follow-up)
  Participants will be asked to tap their right index finger on a standard QWERTY keyboard "1" key when a visual cue appears. The response time for tapping the "1" key, in response to seeing the visual cue, will be measured to assess motor-timing control. Accuracy of response will be dependent on minimizing early or delayed taps (measured in milliseconds) in congruence with the determined rhythm. A change in score, particularly greater accuracy in timing, from baseline indicates better or improved motor control performance.
Change in Continuous Finger Motor Control Timing Abilities from baseline | Week 0 (baseline), week 4 (during), week 8 (end), and week 12 (follow-up)
  Participants will be asked to tap their right index finger on a standard QWERTY keyboard "1" key when a visual cue appears. The participants will then be asked to maintain the tapping rhythm without the visual cue for 15 seconds. The timing of tapping the "1" key, without the visual cue, will be measured to assess motor-timing control. Accuracy of response will be dependent on minimizing early or delayed taps (measured in milliseconds) in congruence with the determined rhythm. A change in score, particularly greater accuracy in timing, from baseline indicates better or improved motor control performance.
Change in Unified Parkinson Disease Rating Scale (UPDRS) from baseline | Week 0 (baseline), week 4 (during), week 8 (end), and week 12 (follow-up)
  UPDRS objectively assesses the severity of PD based off the disease's burden on the individual and can describe disease progression and treatment response. A total of 42 ratings are split between multiple categories. Examples of categories measured include mental impairments (mood and intelligence), activities in daily living (speech, salivation, level of independence to perform normal tasks such as turning in bed), motor skills (facial, tremor severity in extremities, rigidity) and other complications. Each category has a 0-4 rating determined by the examiner and summed, where a higher score reflects greater disability (maxed at 195 points). A change in the score, i.e. lower score from baseline, indicates beneficial effects of the intervention.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Week 0 (baseline), week 4 (during), week 8 (end), and week 12 (follow-up)
  MoCA assesses for an individual's cognitive abilities including orientation, concentration and attention, executive functions, memory, conceptual thinking, calculations, language, and visuo-constructional skills. The test is administered for 10-minutes as a one-page 30-point test. The point distribution is as follows. A short-term memory recall task with five nouns and delayed recall after five minutes (5 points). A clock drawing task (3 points) and a three-dimensional cube copy (1 point) are used to assess visuospatial abilities. Executive functioning is measured using the Trail Making B task (1 point), a phonemic fluency task (1 point), and a two-item abstraction task (2 points). A three-item confrontation naming task (3 points) as well as repeating two sentences with complex syntax (2 points) are used to measure language. Lastly, time and place orientation (6 points) is assessed. A larger total score (> or = 26 is normal) indicates healthy or normal cognition.
n-Back Working Memory Assessment | Week 0 (baseline), week 4 (during), week 8 (end), and week 12 (follow-up)
  The n-back task examines an individual's working memory and working memory capacity by employing a visuo-spatial continuous performance task. This study will use 3-back tasks that are delivered digitally and started with a digital countdown. The participant is asked to input a keystroke on standard QWERTY keyboard with their right-hand to indicate whether a target visual stimulus presented on the screen was identical to a previously shown stimulus presented 'n' trials ago. The stimulus will be a white square randomized into one of six positions on a black screen. The first cue stimulus will be presented on the screen for 3 s and the individual has 3 s to respond with a '1' keystroke to indicate 'same' or a '2' keystroke to indicate 'different'. A new stimulus will appear after a 1 s inter-stimulus interval. Each task will include responses to two sets of 15 and thus each assessment will last approximately 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanhua Liang, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Bingwei Zhang, MD, Principal Investigator — The First Affiliated Hospital of Dalian Medical University; Fengyu Cong, PhD, Principal Investigator — Dalian University of Technology; William C Tang, PhD, Principal Investigator — University of California, Irvine
Locations (1):
- First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pu L, Qureshi NK, Ly J, Zhang B, Cong F, Tang WC, Liang Z. Therapeutic benefits of music-based synchronous finger tapping in Parkinson's disease-an fNIRS study protocol for randomized controlled trial in Dalian, China. Trials. 2020 Oct 16;21(1):864. doi: 10.1186/s13063-020-04770-9. PMID 33066811